CLINICAL TRIAL: NCT03780296
Title: Implementing Technology Enhanced Real Time Action Observation Therapy in Persons With Chronic Stroke
Acronym: TERTAOT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Collaborators: University of Michigan-Flint (Unknown)
Responsible Party: Principal Investigator, Mary Roberts, Physical Therapist, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: HUM00121813
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Last update posted 2018-12-19 (Actual); Status verified 2018-12

CONDITIONS: Chronic Stroke; Hemiplegia; Hemiparesis; Paralysis
Keywords: Kinect; Rehabilitation; Virtual reality; Mirror therapy
MeSH Terms: conditions — Hemiplegia; Paresis; Paralysis

STUDY DESIGN:
Intervention Model Description: Single group pre-test/post-test design
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Real-Time Action Observation with augmented Kinect (Experimental): Participants will receive 30 minutes of the augmented kinect software in real-time undergoing an exercise protocol involving seated upper extremity exercises, seated lower extremity exercises and standing upper extremity exercises.
  Interventions: Device: Real-time action observation with augmented Kinect

INTERVENTIONS:
Device: Real-time action observation with augmented Kinect — Participants will receive 30 minutes of the augmented kinect software in real-time undergoing an exercise protocol involving seated upper extremity exercises, seated lower extremity exercises and standing upper extremity exercises.

SUMMARY:
This is a feasibility study to alter the Microsoft Kinect software to be used as a rehabilitation tool. The prototype used is still in the early developing stage. The purpose of this research study is to develop a prototype of altered Microsoft Kinect Software and determine its use in improving the function of the study subjects' weaker extremities. The altered software will allow a viewing of the mirror image of the involved limb as it is moved. However, the image that is viewed will reflect normal movement even if the limb cannot move normally. By viewing normal movement of the weaker limbs the "mirror neuron" network in the brain will become activated and will ultimately improve the function of the weaker side.

ELIGIBILITY:
Inclusion Criteria:

* - Adults 40 years of age and older having had a stroke greater than 6-months post onset
* Able to follow commands in English
* Medically stable and without acute illness, such as infection, inflammation, ongoing chest pain, or short of breath with walking and light activities
* Able to stand up off of a standard height chair (16-18 inches)

Exclusion Criteria:

* - Cognitive impairment as measured by a score below 24/30 on Mini Mental State Examination
* A diagnoses of cancer involving the nervous or musculoskeletal system
* Severe pain in arms, legs, or spine measured by >6/10 using Verbal Numerical Pain Rating Scale that prevents them from standing or walking independently
* Diagnoses of other neurological diseases except for stroke, such as spinal cord injury or Parkinson's disease etc.
* Individuals at the advanced stage of a disease and with less than 12 months to live.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2017-09-05 (Actual); Primary Completion 2018-09-26 (Actual); Study Completion 2018-09-26 (Actual)

PRIMARY OUTCOMES:
Change in Motor Activity Log (MAL) | 5 months
  MAL measures participants overall use or increased use and quality of use of affected upper limb
Change in 9 Hole Peg Test (9HPT) | 5 months
  9 HPT is a timed standardized measure participants overall function of dexterity.
Change in 10 Meter Walk Test (10mWT) | 5 months
  The 10mWT is a standardized measure used to assess participants timed walking speed in meters per second over a short distance
Change in Functional Reach Test (FRT) | 5 months
  The functional reach test is a standardized measure assessing the participants ability to reach forward with unaffected arm
Change in Timed Up and Go (TUG) | 5 months
  The TUG is a standardized measure which assesses participants mobility, balance, walking ability, and fall risk in older adults
Change in 5 Time Sit to Stand (5xSS) | 5 months
  This is a standardized measure assessing participants functional lower limb strength.

CONTACTS AND LOCATIONS:
Overall Officials: Hendrika L Lietz, PT, DPT, NCS, Study Chair — Michigan Medicine
Locations (1):
- MedRehab Canton, Canton, Michigan, United States

IPD SHARING:
Plan to Share IPD: Yes
Dissemination at local, state and national conferences via platform and poster presentations.
  Share upon request.
Supporting Information: Study Protocol, SAP